CLINICAL TRIAL: NCT04844749
Title: VERACITY - Randomized, Active-Controlled, Phase 3 Study of VERU-111 for the Treatment of Metastatic Castration-Resistant Prostate Cancer in Patients Who Have Failed Prior Treatment With at Least One Androgen Receptor Targeting Agent
Brief Title: Efficacy Evaluation of VERU-111 for mCRPC in Patients Who Have Failed at Least One Androgen Receptor Targeting Agent
Acronym: VERACITY
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Administrative reasons
Sponsor: Veru Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: V3011102
Record Dates: First submitted 2021-04-09; First posted 2021-04-14 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Metastatic Castration-resistant Prostate Cancer; Androgen Resistant Prostatic Cancer
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant | interventions — sabizabulin; enzalutamide; abiraterone; Abiraterone Acetate

STUDY DESIGN:
Intervention Model Description: This randomized, open-label, active-control clinical study consists of two treatment arms:VERU-111 (Sabizabulin) treated group, and Control treated group. Subjects will be randomized in a 2:1 fashion.
Who Masked: Outcomes Assessor
Masking Description: Central reader for scans will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Either VERU-111 32mg or 26mg dose will be supplied as capsules 1 orally once a day (Experimental): 32mg of VERU-111 26mg of VERU-11
  Interventions: Drug: VERU-111
- Active control alternative androgen receptor targeting agent (Active Comparator): The alternative androgen receptor targeting agent will be administered according to the dosing instructions in the current product prescribing information.
  Interventions: Drug: Enzalutamide, Abiraterone

INTERVENTIONS:
Drug: VERU-111 — Based on the safety and antitumor activity of VERU-111 in the Phase 1b/2 clinical study, VERU-111 is initiating this Phase 3 clinical study of VERU-111 for the treatment of metastatic castration resistant prostate cancer in patients who have failed prior treatment with at least one androgen receptor targeting agent
  Other Names: Sabizabulin
  Arms: Either VERU-111 32mg or 26mg dose will be supplied as capsules 1 orally once a day
Drug: Enzalutamide, Abiraterone — Enzalutamide and abiraterone were chosen as active comparators are both are FDA approved for the treatment of metastatic castration resistant prostate cancer
  Other Names: XTANDI; Zytiga
  Arms: Active control alternative androgen receptor targeting agent

SUMMARY:
To demonstrate the efficacy of VERU-111 (Sabizabulin) in the treatment of metastatic castration-resistant prostate cancer in patients who have failed prior treatment with at least one androgen receptor targeting agent as measured by radiographic progression-free survival.

DETAILED DESCRIPTION:
This study is a multicenter, randomized, open-label, active-control, efficacy and safety study of VERU-111 (Sabizabulin) for the treatment of metastatic castration-resistant prostate cancer in patients who have failed prior treatment with at least one androgen receptor targeting agent.

Subjects will have failed treatment with at least one prior androgen receptor targeting agent and be eligible for treatment with an alternative androgen receptor targeting agent (as per the current standard of care for these patients).

Subjects will be randomized in a 2:1 ratio to receive VERU-111 or Active Control (alternative androgen receptor targeting agent).

Subjects in the VERU-111 treated group will receive VERU-111 32 mg per day orally with an option to reduce the dose to 26 mg per day based on tolerability to the 32 mg dose until radiographic progression (blinded independent central read) in observed. Subjects in the Control treated group will receive an alternative androgen receptor targeting agent with dose and dosing regimen defined in the FDA approved prescribing information until radiographic progression in observed.

Randomization will be stratified by measurable disease vs. bone-only disease. A significant proportion (>30%) of the patients randomized into the study will have measurable disease at baseline.

Randomization will also be stratified by if the patient has failed one vs. more than one prior androgen targeting agent.

The primary efficacy endpoint of the study will be radiographic progression free survival.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent.
* Be able to communicate effectively with the study personnel.
* Aged ≥18 years.
* Histological or cytologic proof of adenocarcinoma of the prostate not including the diagnosis of small cell carcinoma of the prostate of neuroendocrine pathology.
* Radiographic evidence of metastatic disease at baseline by CT scan, or MRI and bone scan, with confirmation of measurable disease by RECIST 1.1 and/or identifiable discrete bone metastases by PCWG3.
* Known castration resistant prostate cancer, defined according to PCWG3 criteria.
* Have received at least one androgen receptor targeting agent (e.g. abiraterone, enzalutamide, darolutamide, or apalutamide).
* Subjects who have metastatic castration resistant prostate cancer that have maintained or have previously been treated with ADT (while on-study, patients must receive continuous ADT. Either chemical or surgical castration by bilateral orchiectomy is acceptable) and have failed prior treatment with at least one androgen receptor targeting agent (e.g. abiraterone, enzalutamide, darolutamide, or apalutamide) defined as:
* Serum PSA progression of two consecutive increases in PSA over a previous reference value within 6 months of first study treatment, each measurement at least 2 weeks apart. Or
* Documented bone lesions by the appearance of two or more new lesions on bone scintigraphy or bi-dimensionally-measurable soft tissue metastatic lesion assessed by CT or MRI.
* Treatment with an alternative androgen receptor targeting agent is a reasonable next line of therapy.
* Absolute PSA ≥2.0 ng/ml at screening.
* ECOG performance status <2.
* Participants must have normal organ and bone marrow function measured within 30 days prior to administration of study treatment as defined below:
* Hemoglobin ≥9.0 g/dL with no blood transfusion in the past 30 days
* Creatinine clearance ≥60 mL/min (using Cockcroft-Gault equation)
* Absolute neutrophil count (ANC) ≥1.5 x 109/L
* Platelet count ≥100 x 109/L
* Total bilirubin ≤ upper limit of normal (ULN) (or <2.5 x ULN for patients with known Gilberts disease)
* Aspartate aminotransferase (AST) (Serum Glutamic Oxaloacetic Transaminase (SGOT))/Alanine aminotransferase (ALT) (Serum Glutamic Pyruvate Transaminase (SGPT)) ≤2.5 x ULN. NOTE: Patients with elevations in bilirubin, AST, or ALT should be thoroughly evaluated for the etiology of this abnormality prior to entry and patients with evidence of viral infection should be excluded. Patients with chronic renal stent and stable creatinine elevation can be included in the study with written documentation from the PI.
* Participants must have a life expectancy >3 months.
* Subjects must agree to use acceptable methods of contraception:
* If the study subject's partner could become pregnant, use acceptable methods of contraception from the time of the first administration of study medication until 6months following administration of the last dose of study medication. Acceptable methods of contraception are as follows: Condom with spermicidal foam/gel/film/cream/suppository [i.e.,barrier method of contraception], surgical sterilization (vasectomy with documentation of azospermia) and a barrier method {condom used with spermicidal foam/gel/film/cream/suppository}, the female partner uses oral contraceptives (combination estrogen/progesterone pills), injectable progesterone or subdermal implants and a barrier method (condom used with spermicidal foam/gel/film/cream/suppository).
* If female partner of a study subject has undergone documented tubal ligation (female sterilization), a barrier method (condom used with spermicidal foam/gel/film/cream/suppository)should also be used.-If female partner of a study subject has undergone documented placement of an intrauterine device (IUD) or intrauterine system (IUS),a barrier method (condom with spermicidal foam/gel/film/cream/suppository)should also be used.
* Other than metastatic prostate cancer, no evidence (within 5 years) of prior malignancies (except successfully treated basal cell or squamous cell carcinoma of the skin or other cancers treated with curative intent >3 years prior).
* Participants must agree to refrain from prolonged exposure to the sun or agree to use at least SPF 50 on all exposed skin and protective clothing during prolonged sun exposure throughout participation in this study and/or treatment with VERU- 111.
* Subject is willing to comply with the requirements of the protocol through the end of the study.

Exclusion Criteria:

* Known hypersensitivity or allergy to colchicine.
* Histologic identification of small cell carcinoma of the prostate or neuroendocrine pathology in either biopsy or prostatectomy tissue.
* A bone scan with evidence of superscan or superscan phenomenon, defined as:
* Uptake throughout the axial skeleton and proximal appendicular skeleton, often somewhat heterogeneous, or,
* Symmetrically intense and diffuse radiotracer uptake in the skeleton with absent or diminished visualization of the genitourinary system and soft tissues, or,
* Defined in the bone scan report as a superscan or superscan phenomenon. NOTE: Medical Monitor should be consulted prior to screening of a patient if a superscan or superscan phenomenon is suspected or possible, but undetermined by any of the above definitions.
* Has received external-beam radiotherapy within the last 2 weeks prior to start of study treatment.
* Patients with a QT interval corrected by Fridericia's formula of >480 ms.
* Patients receiving full dose warfarin therapy are not eligible for study.
* Patients with prior history of a thromboembolic event within the last 6 months.
* Participation in another clinical study with an investigational product during the last 6 months prior to randomization into this study.
* Patients should be excluded if they have had prior systemic treatment with prior taxane chemotherapies (for greater than 2 cycles) for advanced prostate cancer. Patient can have up to 2 cycles of prior taxane chemotherapy greater than one year prior to randomization and remain eligible for inclusion in this study. Taxane exposure in the adjuvant or neoadjuvant setting is allowed (maximum of 6 cycles).
* Any treatment modalities involving major surgery within 4weeks prior to the start of study treatment.
* Patients are excluded if they have known brain metastases or leptomeningeal metastases.
* Patients should be excluded if they have a positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection.
* Has imminent or established spinal cord compression based on clinical findings and/or MRI.
* Any other serious illness or medical condition that would, in the opinion of the investigator, make this protocol unreasonably hazardous. Active infections discovered during screening period must be treated and controlled before patient is dosed with VERU-111.
* Persistent toxicities (>Common Terminology Criteria for Adverse Event (CTCAE) grade 2) caused by previous cancer therapy, excluding alopecia.
* Poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 6 months) myocardial infarction, uncontrolled major seizure disorder, extensive interstitial bilateral lung disease, or any psychiatric disorder that prohibits obtaining informed consent.
* Total bilirubin levels > 1.5 x ULN (>2.5 x ULN in patients with known Gilbert's disease).
* AST and/or ALT levels >2.5xULN or AST and/or ALT levels >1.5xULN WITH concomitant alkaline phosphatase levels >2.5xULN.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 105 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-05-04 (Actual)

PRIMARY OUTCOMES:
Efficacy of VERU-111 in the treatment of metastatic castration-resistant prostate cancer in patients who have failed prior treatment with at least one androgen receptor targeting agent | 360 days
  Radiographic progression-free survival (rPFS) centrally read, which is death or tumor progression as defined by RECIST 1.1 (soft tissue) and PCWG3 (bone).

SECONDARY OUTCOMES:
Overall Survival | 360 days
  Overall survival (OS) will be an assessment of time from randomization into the study to all-cause mortality. The analysis will be performed similarly to the primary endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Barnette, Study Chair — Veru Inc.
Locations (40):
- United States (40):
  - Alaska Oncology and Hematology, LLC., Anchorage, Alaska
  - Urology Associates of Southern Arizona, Tucson, Arizona
  - Arizona Urology Specialists, Tucson, Arizona
  - Tower Urology, Los Angeles, California
  - University of California, Irvine, Orange, California
  - West Coaster Center Urology, Oxnard, California
  - San Bernardino Urological Associates, San Bernardino, California
  - Genesis Resaerch, LLC, San Diego, California
  - Genesis Healthcare Partners - Genesis Research Greater Los Angeles, Sherman Oaks, California
  - Alicia Buenrostro, Torrance, California
  - Colorado Urology, Golden, Colorado
  - Universal Axon Clinical Research, Doral, Florida
  - Demirra Hudge, Miami Beach, Florida
  - Florida Urology Partners, LLC, Riverview, Florida
  - Georgia Urology, Atlanta, Georgia
  - Comprehensive Urologic Care, Lake Barrington, Illinois
  - First Urology, PSC, Jeffersonville, Indiana
  - MidAmerica Cancer Care, Merriam, Kansas
  - Chesapeake Urology Research Associates, Baltimore, Maryland
  - Michigan Institute of Urology, Troy, Michigan
  - GU Research Network, LLC, Omaha, Nebraska
  - Inpsira Medical Center Mullica Hill, Mullica Hill, New Jersey
  - Ascension - Our Lady of Lourdes Memorial Hospital, Binghamton, New York
  - Premier Medical Group of the Hudson Valley, Poughkeepsie, New York
  - Associated Medical Professionals of NY, PLCC, Syracuse, New York
  - Associated Urologists of North Carolina, Raleigh, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Clinical Research Solutions - Cleveland, Middleburg Heights, Ohio
  - Oregon Urology Institute, Springfield, Oregon
  - Centers for Advanced Urology, LLP MidLantic Urology, Bala-Cynwyd, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Lexington Medical Center/ Lexington Oncology, West Columbia, South Carolina
  - Urology Associates - Nashville, Nashville, Tennessee
  - Houston Metro Urology, Houston, Texas
  - Urology San Antonio P.A., San Antonio, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Virginia Urology, Richmond, Virginia
  - Urology of Virginia, PLLC, Virginia Beach, Virginia
  - Spokane Urology P.S., Spokane, Washington
  - Cancer Care Northwest, Spokane Valley, Washington

IPD SHARING:
Plan to Share IPD: No